CLINICAL TRIAL: NCT02652585
Title: Validation of a Test System for Development of Medications for Alcoholism
Acronym: TEMANX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: TUD-TEMANX-065
Record Dates: First submitted 2016-01-06; First posted 2016-01-12 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Alcoholism
Keywords: Alcoholism; alcohol self-administration
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naltrexone (Active Comparator): 1 capsule naltrexone 25 mg per day, oral use, day 1 to day 3;
  1 capsule naltrexone 50 mg per day, oral use, day 4 to day 28
  Interventions: Drug: Naltrexone
- Placebo (Placebo Comparator): 1 capsule placebo, oral use, day 1 to day 28
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone
  Other Names: Adepend
  Arms: Naltrexone
Drug: Placebo — capsule filled with micro crystalline cellulose, manufactured to mimic naltrexone capsule
  Arms: Placebo

SUMMARY:
Using theTEMA (test system for development of medications for alcoholism) it can be shown, that naltrexone administration reduces the willingness to perform work for alcohol infusion in a laboratory experiment.

DETAILED DESCRIPTION:
Objective of this study is to show that a laboratory alcohol self-administration method can predict the therapeutic potential of new compounds to reduce relapse in alcohol-dependent patients.

The 'TEMA" translates several animal behavioral paradigms of alcohol self-administration into corresponding human experiments.

We will investigate the opiate antagonist Naltrexone, whose anti-relapse effect is well documented, as a reference drug for validation.

Main objective:

With TEMA (test system for development of medications for alcoholism ) it can be shown, that naltrexone administration reduces the willingness to perform work for alcohol infusion in a laboratory experiment.

Secondary objectives:

* administration of naltrexone in comparison to placebo leads to a reduction of alcohol craving and real-life drinking
* administration of naltrexone in comparison to placebo leads to reduction of the CDT-Level
* administration of naltrexone in comparison to placebo leads to a change in perception of subjective alcohol effects
* the effectiveness of naltrexone can be predicted by the A118G polymorphism of the OPRM1
* administration of naltrexone changes the baseline and alcohol-induced ability of motor inhibition
* administration of naltrexone changes the baseline and alcohol-induced regional cerebral perfusion
* administration of naltrexone changes the baseline and alcohol-induced cerebral resting state activity
* changes of alcohol effects to the brain activity induced by naltrexone in comparison to placebo correlate with effects of naltrexone on the willingness to work for alcohol self-administration

ELIGIBILITY:
Inclusion Criteria:

* male and female volunteers aged 25 to 55 years
* at least weekly alcohol consumption at a medium risk level according to WHO in the Timeline Follow-back Interview over the last 45 day with an average amount of alcohol of 41 g/day (men) or 31 g/day (women)
* at least 6 days with an alcohol consumption of >100 g/day (men) or 75 g/day (women) and at least 4 non consecutive alcohol abstinent days in the last 45 days
* at least 1 drinking day in each full week between screening and visit 1 and not more than 6 abstinent days in the week before visit 1
* no demand of treatment of the risky alcohol consumption
* written consent after Information

Exclusion Criteria:

* a history of hypersensitivity against alcohol or one of the used medicinal products, of their ingredients or medicinal products with similar chemical structures
* participation in another clinical trial within the last 4 weeks before inclusion
* addiction or other disorders, which will not allow the subject to assess the character and importance or possible consequences of the clinical trial
* pregnant or breastfeeding women
* women capable of bearing children, except women who fulfil following criteria:- post-menopausal (12 months natural amenorrhoea or 6 month amenorrhoea and Serum FSH >40 ml U/ml) - post operative (6 weeks after ovariectomy on both sides with or without hysterectomy) - regular and correct use of a contraceptive method with an error Quote of < 1 % per year (for example implants, depot injections, oral contraceptive, IUP). It has to be recognized that a combined oral contraception - in contrast to pure progesterone compounds - have a failure rate of < 1 %. Hormone IUDs with a Pearl Index of 1 % are safer than copper IUDs. - sexual abstinence - vasectomy of the Partner
* evidence that the participant is not expected to comply with the protocol (for example lacking compliance)
* current or previous alcohol or substance dependence according to DSM-IV (exception: tobacco dependence)
* current or previous treatment because of alcohol, for example in an addiction advisory cen-tre, self-help group, detoxification treatment
* current or previous diseases, where an alcohol infusion can cause a clinically relevant hazard (e. g. pancreatitis, liver cirrhosis)
* current or planned intake of opiate analgesics
* current psychiatric treatment or intake of psychiatric drug or suffering from of a psychiatric disease requiring treatment
* a history of suicide attempt
* CIWA-Score >5 at Screening (alcohol withdrawal scale)
* a history of symptoms of alcohol withdrawal, epileptic seizures or delirium
* routine laboratory Parameters, indicating relevant liver-, pancreas- or kidney injury, an acute infection, anaemia or lack of vitamins (ASAT, ALAT > twofold of the standard at screening, gamma-GT, lipase >threefold of the standard, CRP < 15 mg/l, creatin indicating a moderate renal insufficiency ( eGFR <60 ml/min), leucocytes > 12000/µl, haemoglobin < 7,5 mmol/l (men) or 6,5 mmol/l (women), MCV > 100 fl)
* Body weight > 130 kg
* drug screening in urine: once positive at screening for opiate, cannabis, cocaine, amphetamines, benzodiazepines or positive once at visit 1 for opiates or positive twice at visit 1 for cannabis, cocaine, amphetamines, benzodiazepines
* breath alcohol concentration at screening once > 0,00 g/kg or twice >0,00 g/kg at visit 1
* unsuitable for fMRT (e. g. cardiac pacemaker, claustrophobia)
* specific contraindications against naltrexone: o acute hepatitis o severe or acute liver disease o severe kidney disease o rare hereditary galactose intolerance, Lapp-lactase-deficiency or Glucose-galactose-malabsorption

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2017-09-04 (Actual)

PRIMARY OUTCOMES:
Difference CAT Trials alcohol | one year
  Difference of cumulative number of work sets for alcohol in the "constant attention task" between first measurement (without medication) and second measurement (with medication)

SECONDARY OUTCOMES:
Difference CAT Trials sodium chloride solution | one year
  Difference of cumulative number of work sets for sodium chloride solution in the "constant attention task" between first measurement (without medication) and second measurement (with medication)
break Point alcohol | one year
  Difference of the "break point" in the "progressive work" schedule for the work for alcohol between first measurement (without medication) and second measurement (with medication). The "break point" is the number of the last alcohol request before subjects stop to work for more alcohol.
max. BAC | one year
  Maximal achieved blood alcohol concentration (BAC) in alcohol self-administration between first measurement (without medication) and second measurement (with medication)
Drinking habits | one year
  Drinking habits measured with Timeline Follow-back Interview over 45 days before study start (measured at screening) and over the entire study duration (between screening and the last day of medicinal product intake, ascertained at visit 5): drinking days, amount of alcohol per drinking day and number of days with alcohol consumption over 60 g (men) or 48 g (women)
CDT - level | one year
  CDT - level: (carbohydrate-deficient transferrin), measured at visit 1 and visit 5
alcohol craving | one year
  Alcohol craving in daily routine (OCD - scale) measured at visit 1 and visit 4
subjective alcohol effects | one year
  Difference in subjective alcohol effects between first measurement (without medication) and second measurement (with medication), measured with visual analogue scales ("Quizzer") before, during and after the alcohol infusion
motor impulse control | one year
  Capacity for motor impulse control during infusion of physiologic saline solution or alcohol as NIMPs (single-blinded), measured with the counting stroop task (in Verum and placebo group) at visit 3 and 4
cerebral blood flow (CBF) | one year
  Regional cerebral perfusion in ml/100 g tissue per Minute during infusion of sodium chloride solution or alcohol as NIMPs (single-blinded), measured with arterial spin labeling (ASL) under verum or placebo condition at visit 3 and 4
Cerebral resting state activity | one year
  Cerebral resting state activity during infusion of sodium chloride solution or alcohol as NIMPs (single-blinded), measured with BOLD fMRI (in Verum and placebo group) at visit 3 and 4
adverse events | one year
  Medical survey concerning occurring adverse events at visit 1 to 5
ALAT | one year
  ALAT (alanine aminotransferase) in µmol/ s*l before inclusion (screening visit), at visit 4 and after finishing all study relating interventions (visit 5)
ASAT | one year
  ASAT (aspartate aminotransferase) in µmol/ s*l before inclusion (screening visit), at visit 4 and after finishing all study relating interventions (visit 5)
Gamma-GT | one year
  Gamma-GT in µmol/ s*l before inclusion (screening visit) and after finishing all study relating interventions (visit 5)
standard blood cell count | one year
  standard blood cell count before inclusion (screening visit), at visit 4 and after finishing all study relating interventions (visit 5)
creatinine | one year
  creatinine in µmol/l before inclusion (screening visit)
lipase | one year
  lipase in µmol/ s*l before inclusion (screening visit) and after finishing all study relating interventions (visit 5)
CRP | one year
  CRP (C-reactive protein) in mg / l before inclusion (screening visit) and after finishing all study relating interventions (visit 5)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich S Zimmermann, MD, Study Director — Klinik und Poliklinik für Psychiatrie und Psychotherapie Unversitätsklinikum Carl Gustav Carus Dresden
Locations (1):
- Klinik und Poliklinik für Psychiatrie und Psychotherapie, Dresden, Germany

IPD SHARING:
Plan to Share IPD: Undecided